CLINICAL TRIAL: NCT00559754
Title: An Open Label Study to Assess the Effect of a Combination of Avastin and Docetaxel and Sequential Chemotherapy on Pathological Response in Patients With Primary Operable HER2 Negative Breast Cancer
Brief Title: A Study of Avastin (Bevacizumab) and Sequential Chemotherapy in Patients With Primary HER2 Negative Operable Breast Cancer.
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ML20382
Record Dates: First submitted 2007-11-15; First posted 2007-11-16 (Estimated); Results first posted 2014-11-10 (Estimated); Last update posted 2014-11-10 (Estimated); Status verified 2014-11

CONDITIONS: Breast Cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — Bevacizumab; Docetaxel

ARMS (1):
- 1 (Experimental)
  Interventions: Drug: bevacizumab [Avastin]; Drug: Docetaxel; Drug: Standard chemotherapy

INTERVENTIONS:
Drug: bevacizumab [Avastin] — 15mg/kg iv on day 1 of each 3 week cycle
Drug: Docetaxel — 75mg/m2 iv on day 1 of each 3 week cycle
Drug: Standard chemotherapy — As prescribed

SUMMARY:
This single arm study will assess the efficacy and safety of a combination of Avastin and docetaxel following cyclophosphamide and doxorubicin, in patients with HER2 negative operable breast cancer. Patients will receive 4 x 3 week cycles of chemotherapy with doxorubicin (60mg/m2 iv on day 1 of each cycle) and cyclophosphamide (600mg/m2 iv on day 1 of each cycle). They will then receive 4 x 3 week cycles of docetaxel (75mg/m2 on day 1 of each cycle) in combination with Avastin (15mg/kg on day 1 of each cycle). The anticipated time on study treatment is 3-12 months, and the target sample size is <100 individuals.

ELIGIBILITY:
Inclusion Criteria:

* female patients, >=18 years of age;
* primary HER2-negative operable breast cancer;
* tumor >2cm in size;
* ECOG performance status 0-1.

Exclusion Criteria:

* previous treatment for breast cancer;
* metastatic disease;
* current or recent (within 10 days of first dose of Avastin) use of aspirin (>325mg/day) or full-dose anticoagulants for therapeutic purposes;
* clinically significant cardiovascular disease.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 72 (Actual)
Dates: Start 2007-12; Primary Completion 2010-09 (Actual); Study Completion 2010-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (6):
- Spain (6):
  - Sabadell, Barcelona, Barcelona
  - Córdoba, Cordoba
  - Jaén, Jaen
  - Lleida, Lerida
  - Málaga, Malaga
  - Zaragoza, Zaragoza

RESULTS

PARTICIPANT FLOW:
Groups:
- Doxorubicin + Cyclophosphamide/Bevacizumab + Docetaxel: Participants received doxorubicin 60 milligrams per square meter (mg/m^2) intravenously (IV) followed by cyclophosphamide 600 mg/m^2 IV on Day 1, repeated every 3 weeks for a maximum of 4 cycles.
  Participants then received bevacizumab 15 mg per kilogram (mg/kg) IV followed by docetaxel 75 mg/m^2 IV on Day 1, repeated every 3 weeks for a maximum of 4 cycles.
Period: Overall Study
Arm/Group | Doxorubicin + Cyclophosphamide/Bevacizumab + Docetaxel
Started | 72
Completed | 61
Not Completed | 11
Not completed — Disease progression | 1
Not completed — Adverse Event | 5
Not completed — Protocol Violation | 1
Not completed — Investigator criteria | 2
Not completed — Withdrawal by Subject | 2

BASELINE CHARACTERISTICS:
Population: Intent to Treat (ITT) Population: all participants included in the study.
Groups:
- Doxorubicin + Cyclophosphamide/Bevacizumab + Docetaxel: Participants received doxorubicin 60 mg/m^2 IV followed by cyclophosphamide 600 mg/m^2 IV on Day 1, repeated every 3 weeks for a maximum of 4 cycles. Participants then received bevacizumab 15 mg/kg IV followed by docetaxel 75 mg/m^2 IV on Day 1, repeated every 3 weeks for a maximum of 4 cycles.
Arm/Group | Doxorubicin + Cyclophosphamide/Bevacizumab + Docetaxel
Number analyzed (Participants) | 72
Age, Continuous [Mean (Standard Deviation); unit: years] | 47.22 (9.85)
Sex/Gender, Customized [Number; unit: participants]
  Female | 72

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Pathological Complete Response (pCR)
Description: The percentage of participants with pCR was determined by anatomopathological study after completion of 8 cycles of study treatment. The anatomopathological study of the surgical piece was performed and assessed according to the Miller-Payne criteria: 1) the primary tumor was Grade 5 (no malignant cells identified at the location of the primary tumor (ductal carcinoma in situ may be present); 2) no involvement was identified in the lymph nodes; 3) the tumour size at evaluation of the surgical piece was 0 centimeters (cm); and 4) the pathological staging of the tumour from the surgical piece was pT0pN0pM0, the stage is not applicable (NA). It will only be considered pCR in the case of absence of invasive tumour cells in the breast and lymph nodes.
Time Frame: After Week 24 (surgery)
Population: Population evaluable for anatomopathological response: participants who satisfied all inclusion criteria and none of the exclusion criteria, received at least 2 cycles of chemotherapy treatment, and were evaluated pathologically.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Doxorubicin + Cyclophosphamide/Bevacizumab + Docetaxel
Number analyzed (Participants) | 66
percentage of participants | 24.2 [14.5 to 36.4]

2. Secondary Outcome: Percentage of Participants With Objective Clinical Response
Description: Overall clinical response is the best response obtained through physical examination and/or radiological tests after completion of chemotherapy cycles. The percentage of participants with objective response based on assessment of complete response (CR) or partial response (PR) according to Response Evaluation Criteria in Solid Tumors (RECIST) and was categorized as clinical response (CR+PR) or clinical benefit (CR+PR+ no change [NC]). Per RECIST, CR was defined as disappearance of all target lesions, non-target lesions, and normalization of tumor marker level. PR was defined as greater than or equal to (≥)30 percent (%) decrease under baseline of the sum of the longest diameter (LD) of all target lesions. No unequivocal progression of non-target disease. No new lesions. Complete and partial responses must have been confirmed no less than 4 weeks after the criteria for response were first met.
Time Frame: Within 28 days of enrollment, Weeks 12 and 24
Population: ITT Population
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Doxorubicin + Cyclophosphamide/Bevacizumab + Docetaxel
Number analyzed (Participants) | 72
percentage of participants
  CR+PR | 88.9 [79.3 to 95.1]
  CR+PR+NC | 98.6 [92.5 to 99.9]

3. Secondary Outcome: Percentage of Participants With Breast-Conserving Surgery
Description: Breast-conserving surgery was defined as lumpectomy + lymphadenectomy (LA), segmentectomy + LA, quadrantectomy + LA, or other (including sentinal node extirpation tumorectomy).
Time Frame: Week 24
Population: ITT population; only those participants who underwent surgery were included in the analysis
Measure: Number; unit: percentage of participants
Arm/Group | Doxorubicin + Cyclophosphamide/Bevacizumab + Docetaxel
Number analyzed (Participants) | 67
percentage of participants | 62.7

4. Secondary Outcome: Percentage of Participants With pCR by Proliferation of Ki67
Description: The percentage of participants with pCR was determined by anatomopathological study after completion of 8 cycles of study treatment. The anatomopathological study of the surgical piece was performed and assessed according to the Miller-Payne criteria. It was only considered pCR in the case of absence of invasive tumour cells in the breast and lymph nodes. Biomarker Ki67 proliferation was defined as low (less than [<]15% ) and high (≥15%).
Time Frame: After Week 24 (surgery)
Population: Population evaluable for anatomopathological response with evaluable levels of the specified biomarker; data were missing for 2 participants.
Measure: Number; unit: percentage of participants
Arm/Group | Doxorubicin + Cyclophosphamide/Bevacizumab + Docetaxel
Number analyzed (Participants) | 65
percentage of participants
  High proliferative index (n=50) | 24.0
  Low proliferative index (n=15) | 13.3
Statistical Analysis 1: Comparison: Doxorubicin + Cyclophosphamide/Bevacizumab + Docetaxel; Test type: Superiority or Other; p = 0.4915, Fisher Exact

5. Secondary Outcome: Percentage of Participants With pCR by Kisspeptin (KISS1) Amplification
Description: The percentage of participants with pCR was determined by anatomopathological study after completion of 8 cycles of study treatment. The anatomopathological study of the surgical piece was performed and assessed according to the Miller-Payne criteria. It was only considered pCR in the case of absence of invasive tumour cells in the breast and lymph nodes. KISS1 amplification was defined as 1 (aneuploid), 2 (normal), 4 (amplification), or NE (not evaluated).
Time Frame: After Week 24 (surgery)
Population: Only those participants evaluated for the specified biomarker were included in the analysis.
Measure: Number; unit: percentage of participants
Arm/Group | Doxorubicin + Cyclophosphamide/Bevacizumab + Docetaxel
Number analyzed (Participants) | 23
percentage of participants
  Anueploid (n=8) | 12.5
  Normal (n=13) | 30.77
  Amplification (n=2) | 50.0
Statistical Analysis 1: Comparison: Doxorubicin + Cyclophosphamide/Bevacizumab + Docetaxel; Test type: Superiority or Other; p = 0.4864, Chi-squared

6. Secondary Outcome: Percentage of Participants With pCR by KISS1 Protein Expression
Description: The percentage of participants with pCR was determined by anatomopathological study after completion of 8 cycles of study treatment. The anatomopathological study of the surgical piece was performed and assessed according to the Miller-Payne criteria. It was only considered pCR in the case of absence of invasive tumour cells in the breast and lymph nodes. KISS1 protein expression was defined as 0 (no expression), 1 (normal), 2 (augmented expression), or NE (not evaluated).
Time Frame: After Week 24 (surgery)
Population: Only those participants evaluated for the specified biomarker were included in the analysis.
Measure: Number; unit: percentage of participants
Arm/Group | Doxorubicin + Cyclophosphamide/Bevacizumab + Docetaxel
Number analyzed (Participants) | 25
percentage of participants
  No expression (n=18) | 27.8
  Normal (n=3) | 66.7
  Augmented expression (n=4) | 50.0
Statistical Analysis 1: Comparison: Doxorubicin + Cyclophosphamide/Bevacizumab + Docetaxel; Test type: Superiority or Other; p = 0.3613, Fisher Exact

7. Secondary Outcome: Percentage of Participants With pCR by Vascular Endothelial Growth Factor Receptor (VEGFR) Amplification
Description: The percentage of participants with pCR was determined by anatomopathological study after completion of 8 cycles of study treatment. The anatomopathological study of the surgical piece was performed and assessed according to the Miller-Payne criteria. It was only considered pCR in the case of absence of invasive tumour cells in the breast and lymph nodes. VEFGR amplification was defined as 1 (aneuploid), 2 (normal), 4 (amplification), or NE (not evaluated).
Time Frame: After Week 24 (surgery)
Population: Only those participants evaluated for the specified biomarker were included in the analysis.
Measure: Number; unit: percentage of participants
Arm/Group | Doxorubicin + Cyclophosphamide/Bevacizumab + Docetaxel
Number analyzed (Participants) | 23
percentage of participants
  Anueploid (n=1) | 0
  Normal (n=18) | 33.3
  Amplification (n=4) | 0
Statistical Analysis 1: Comparison: Doxorubicin + Cyclophosphamide/Bevacizumab + Docetaxel; Test type: Superiority or Other; p = 0.6605, Fisher Exact

8. Secondary Outcome: Percentage of Participants With pCR by VEGFR Protein Expression
Description: The percentage of participants with pCR was determined by anatomopathological study after completion of 8 cycles of study treatment. The anatomopathological study of the surgical piece was performed and assessed according to the Miller-Payne criteria. It was only considered pCR in the case of absence of invasive tumour cells in the breast and lymph nodes. VEGFR protein expression was defined as 0 (no expression), 1 (normal), 2 (augmented expression), or NE (not evaluated).
Time Frame: After Week 24 (surgery)
Population: Only those participants evaluated for the specified biomarker were included in the analysis.
Measure: Number; unit: percentage of participants
Arm/Group | Doxorubicin + Cyclophosphamide/Bevacizumab + Docetaxel
Number analyzed (Participants) | 22
percentage of participants
  No expression (n=7) | 28.6
  Normal (n=5) | 40.0
  Augmented expression (n=10) | 20.0
Statistical Analysis 1: Comparison: Doxorubicin + Cyclophosphamide/Bevacizumab + Docetaxel; Test type: Superiority or Other; p = 0.8311, Fisher Exact

9. Secondary Outcome: Percentage of Participants With pCR by Hypoxia Inducible Factor (HIF) Protein Expression
Description: The percentage of participants with pCR was determined by anatomopathological study after completion of 8 cycles of study treatment. The anatomopathological study of the surgical piece was performed and assessed according to the Miller-Payne criteria. It was only considered pCR in the case of absence of invasive tumour cells in the breast and lymph nodes. HIF protein expression was defined as 0 (no expression), 1 (normal), 2 (augmented expression), or NE (not evaluated).
Time Frame: After Week 24 (surgery)
Population: Only those participants evaluated for the specified biomarker were included in the analysis.
Measure: Number; unit: percentage of participants
Arm/Group | Doxorubicin + Cyclophosphamide/Bevacizumab + Docetaxel
Number analyzed (Participants) | 38
percentage of participants
  No expression (n=25) | 40.0
  Normal (n=8) | 12.5
  Augmented expression (n=5) | 60.0
Statistical Analysis 1: Comparison: Doxorubicin + Cyclophosphamide/Bevacizumab + Docetaxel; Test type: Superiority or Other; p = 0.2230, Fisher Exact

10. Secondary Outcome: Percentage of Participants With pCR by Endothelial Nitric Oxide Synthase (ENOS) Protein Expression
Description: The percentage of participants with pCR was determined by anatomopathological study after completion of 8 cycles of study treatment. The anatomopathological study of the surgical piece was performed and assessed according to the Miller-Payne criteria. It was only considered pCR in the case of absence of invasive tumour cells in the breast and lymph nodes. ENOS protein expression was defined as 0 (no expression), 1 (normal), 2 (augmented expression), or NE (not evaluated).
Time Frame: After Week 24 (surgery)
Population: Only those participants evaluated for the specified biomarker were included in the analysis.
Measure: Number; unit: percentage of participants
Arm/Group | Doxorubicin + Cyclophosphamide/Bevacizumab + Docetaxel
Number analyzed (Participants) | 38
percentage of participants
  No expression (n=24) | 29.2
  Normal (n=10) | 40.0
  Augmented expression (n=4) | 25.0
Statistical Analysis 1: Comparison: Doxorubicin + Cyclophosphamide/Bevacizumab + Docetaxel; Test type: Superiority or Other; p = 0.8696, Fisher Exact

11. Secondary Outcome: Percentage of Participants With pCR by Angiotension Protein Expression
Description: The percentage of participants with pCR was determined by anatomopathological study after completion of 8 cycles of study treatment. The anatomopathological study of the surgical piece was performed and assessed according to the Miller-Payne criteria. It was only considered pCR in the case of absence of invasive tumour cells in the breast and lymph nodes. Angiotensin protein expression was defined as 0 (no expression), 1 (normal), 2 (augmented expression), or NE (not evaluated).
Time Frame: After Week 24 (surgery)
Population: Only those participants evaluated for the specified biomarker were included in the analysis.
Measure: Number; unit: percentage of participants
Arm/Group | Doxorubicin + Cyclophosphamide/Bevacizumab + Docetaxel
Number analyzed (Participants) | 26
percentage of participants
  No expression (n=14) | 7.1
  Normal (n=1) | 0.0
  Augmented expression (n=11) | 63.6
Statistical Analysis 1: Comparison: Doxorubicin + Cyclophosphamide/Bevacizumab + Docetaxel; Test type: Superiority or Other; p = 0.0074, Fisher Exact

12. Secondary Outcome: Percentage of Participants With pCR by Vascular Endothelial Growth Factor (VEGF) Gene Expression
Description: The percentage of participants with pCR was determined by anatomopathological study after completion of 8 cycles of study treatment. The anatomopathological study of the surgical piece was performed and assessed according to the Miller-Payne criteria. It was only considered pCR in the case of absence of invasive tumour cells in the breast and lymph nodes. VEGF gene expression was defined as below the housekeeping reference level (>0), above the housekeeping reference level (<0), or equal to the housekeeping reference level (0).
Time Frame: After Week 24 (surgery)
Population: Only those participants evaluated for the specified biomarker were included in the analysis.
Measure: Number; unit: percentage of participants
Arm/Group | Doxorubicin + Cyclophosphamide/Bevacizumab + Docetaxel
Number analyzed (Participants) | 34
percentage of participants
  Gene expression above housekeeping level (n=1) | 100.0
  Gene expression below housekeeping level (n=33) | 30.3
Statistical Analysis 1: Comparison: Doxorubicin + Cyclophosphamide/Bevacizumab + Docetaxel; Test type: Superiority or Other; p = 0.3235, Fisher Exact

13. Secondary Outcome: Percentage of Participants With pCR by VEGFR Gene Expression
Description: The percentage of participants with pCR was determined by anatomopathological study after completion of 8 cycles of study treatment. The anatomopathological study of the surgical piece was performed and assessed according to the Miller-Payne criteria. It was only considered pCR in the case of absence of invasive tumour cells in the breast and lymph nodes. VEGFR gene expression was defined as below the housekeeping reference level (>0), above the housekeeping reference level (<0), or equal to the housekeeping reference level (0).
Time Frame: After Week 24 (surgery)
Population: Only those participants evaluated for the specified biomarker were included in the analysis.
Measure: Number; unit: percentage of participants
Arm/Group | Doxorubicin + Cyclophosphamide/Bevacizumab + Docetaxel
Number analyzed (Participants) | 34
percentage of participants
  Gene expression above housekeeping level (n=7) | 0.0
  Gene expression below housekeeping level (n=27) | 40.7
Statistical Analysis 1: Comparison: Doxorubicin + Cyclophosphamide/Bevacizumab + Docetaxel; Test type: Superiority or Other; p = 0.0693, Fisher Exact

14. Secondary Outcome: Percentage of Participants With pCR by Phosphorylated AKT (pAKT) Gene Expression
Description: The percentage of participants with pCR was determined by anatomopathological study after completion of 8 cycles of study treatment. The anatomopathological study of the surgical piece was performed and assessed according to the Miller-Payne criteria. It was only considered pCR in the case of absence of invasive tumour cells in the breast and lymph nodes. pAKT gene expression was defined as below the housekeeping reference level (>0), above the housekeeping reference level (<0), or equal to the housekeeping reference level (0).
Time Frame: After Week 24 (surgery)
Population: Only those participants evaluated for the specified biomarker were included in the analysis.
Measure: Number; unit: percentage of participants
Arm/Group | Doxorubicin + Cyclophosphamide/Bevacizumab + Docetaxel
Number analyzed (Participants) | 34
percentage of participants
  Gene expression above housekeeping level (n=0) | NA — No participants assessed had PAKT gene expression above the housekeeping level.
  Gene expression below housekeeping level (n=34) | 32.4

15. Secondary Outcome: Percentage of Participants With pCR by HIF Gene Expression
Description: The percentage of participants with pCR was determined by anatomopathological study after completion of 8 cycles of study treatment. The anatomopathological study of the surgical piece was performed and assessed according to the Miller-Payne criteria. It was only considered pCR in the case of absence of invasive tumour cells in the breast and lymph nodes. HIF gene expression was defined as below the housekeeping reference level (>0), above the housekeeping reference level (<0), or equal to the housekeeping reference level (0).
Time Frame: After Week 24 (surgery)
Population: Only those participants evaluated for the specified biomarker were included in the analysis.
Measure: Number; unit: percentage of participants
Arm/Group | Doxorubicin + Cyclophosphamide/Bevacizumab + Docetaxel
Number analyzed (Participants) | 34
percentage of participants
  Gene expression above housekeeping level (n=9) | 44.4
  Gene expression below housekeeping level (n=25) | 28.0
Statistical Analysis 1: Comparison: Doxorubicin + Cyclophosphamide/Bevacizumab + Docetaxel; Test type: Superiority or Other; p = 0.4254, Fisher Exact

16. Secondary Outcome: Percentage of Participants With pCR by Insulin-Like Growth Factor (IGF) Gene Expression
Description: The percentage of participants with pCR was determined by anatomopathological study after completion of 8 cycles of study treatment. The anatomopathological study of the surgical piece was performed and assessed according to the Miller-Payne criteria. It was only considered pCR in the case of absence of invasive tumour cells in the breast and lymph nodes. IGF gene expression was defined as below the housekeeping reference level (>0), above the housekeeping reference level (<0), or equal to the housekeeping reference level (0).
Time Frame: After Week 24 (surgery)
Population: Only those participants evaluated for the specified biomarker were included in the analysis.
Measure: Number; unit: percentage of participants
Arm/Group | Doxorubicin + Cyclophosphamide/Bevacizumab + Docetaxel
Number analyzed (Participants) | 34
percentage of participants
  Gene expression above housekeeping level (n=0) | NA — All participants assessed had IGF gene expression levels below the housekeeping level.
  Gene expression below housekeeping level (n=34) | 32.4

17. Secondary Outcome: Percentage of Participants With pCR by ENOS Gene Expression
Description: The percentage of participants with pCR was determined by anatomopathological study after completion of 8 cycles of study treatment. The anatomopathological study of the surgical piece was performed and assessed according to the Miller-Payne criteria. It was only considered pCR in the case of absence of invasive tumour cells in the breast and lymph nodes. ENOS gene expression was defined as below the housekeeping reference level (>0), above the housekeeping reference level (<0), or equal to the housekeeping reference level (0).
Time Frame: After Week 24 (surgery)
Population: Only those participants evaluated for the specified biomarker were included in the analysis.
Measure: Number; unit: percentage of participants
Arm/Group | Doxorubicin + Cyclophosphamide/Bevacizumab + Docetaxel
Number analyzed (Participants) | 34
percentage of participants
  Gene expression above housekeeping level (n=1) | 0
  Gene expression below housekeeping level (n=33) | 33.3
Statistical Analysis 1: Comparison: Doxorubicin + Cyclophosphamide/Bevacizumab + Docetaxel; Test type: Superiority or Other; p = 1.0000, Fisher Exact

18. Secondary Outcome: Percentage of Participants With pCR by Phosphorylated MAP Kinase (pMAPK) Gene Expression
Description: The percentage of participants with pCR was determined by anatomopathological study after completion of 8 cycles of study treatment. The anatomopathological study of the surgical piece was performed and assessed according to the Miller-Payne criteria. It was only considered pCR in the case of absence of invasive tumour cells in the breast and lymph nodes. pMAPK gene expression was defined as below the housekeeping reference level (>0), above the housekeeping reference level (<0), or equal to the housekeeping reference level (0).
Time Frame: After Week 24 (surgery)
Population: Only those participants evaluated for the specified biomarker were included in the analysis.
Measure: Number; unit: percentage of participants
Arm/Group | Doxorubicin + Cyclophosphamide/Bevacizumab + Docetaxel
Number analyzed (Participants) | 34
percentage of participants
  Gene expression above housekeeping level (n=30) | 33.3
  Gene expression equal to housekeeping level (n=1) | 0
  Gene expression below housekeeping level (n=3) | 33.3
Statistical Analysis 1: Comparison: Doxorubicin + Cyclophosphamide/Bevacizumab + Docetaxel; Test type: Superiority or Other; p = 1.0000, Fisher Exact

19. Secondary Outcome: Percentage of Participants With pCR by Angiotensin II Receptor Type I (AGTR) Gene Expression
Description: The percentage of participants with pCR was determined by anatomopathological study after completion of 8 cycles of study treatment. The anatomopathological study of the surgical piece was performed and assessed according to the Miller-Payne criteria. It was only considered pCR in the case of absence of invasive tumour cells in the breast and lymph nodes. AGTR gene expression was defined as below the housekeeping reference level (>0), above the housekeeping reference level (<0), or equal to the housekeeping reference level (0).
Time Frame: After Week 24 (surgery)
Population: Only those participants evaluated for the specified biomarker were included in the analysis.
Measure: Number; unit: percentage of participants
Arm/Group | Doxorubicin + Cyclophosphamide/Bevacizumab + Docetaxel
Number analyzed (Participants) | 33
percentage of participants
  Gene expression above housekeeping level (n=0) | NA — All participants had AGTR gene exptression below the housekeeping level.
  Gene expression below housekeeping level (n=33) | 30.3

20. Secondary Outcome: Percentage of Participants With pCR by KISS1 Gene Expression
Description: The percentage of participants with pCR was determined by anatomopathological study after completion of 8 cycles of study treatment. The anatomopathological study of the surgical piece was performed and assessed according to the Miller-Payne criteria. It was only considered pCR in the case of absence of invasive tumour cells in the breast and lymph nodes. KISS1 gene expression was defined as below the housekeeping reference level (>0), above the housekeeping reference level (<0), or equal to the housekeeping reference level (0).
Time Frame: After Week 24 (surgery)
Population: Only those participants evaluated for the specified biomarker were included in the analysis.
Measure: Number; unit: percentage of participants
Arm/Group | Doxorubicin + Cyclophosphamide/Bevacizumab + Docetaxel
Number analyzed (Participants) | 34
percentage of participants
  Gene expression above housekeeping level (n=1) | 0.0
  Gene expression below housekeeping level (n=33) | 33.3
Statistical Analysis 1: Comparison: Doxorubicin + Cyclophosphamide/Bevacizumab + Docetaxel; Test type: Superiority or Other; p = 1.0000, Fisher Exact

21. Secondary Outcome: Percentage of Participants With pCR by RKISS1 Gene Expression
Description: The percentage of participants with pCR was determined by anatomopathological study after completion of 8 cycles of study treatment. The anatomopathological study of the surgical piece was performed and assessed according to the Miller-Payne criteria. It was only considered pCR in the case of absence of invasive tumour cells in the breast and lymph nodes. RKISS1 gene expression was defined as below the housekeeping reference level (>0), above the housekeeping reference level (<0), or equal to the housekeeping reference level (0).
Time Frame: After Week 24 (surgery)
Population: Only those participants evaluated for the specified biomarker were included in the analysis.
Measure: Number; unit: percentage of participants
Arm/Group | Doxorubicin + Cyclophosphamide/Bevacizumab + Docetaxel
Number analyzed (Participants) | 34
percentage of participants
  Gene expression above housekeeping level (n=0) | NA — All participants had RKISS1 gene expression below the housekeeping level.
  Gene expression below housekeeping level (n=34) | 32.4

ADVERSE EVENTS:
Time Frame: Adverse events (AEs) were reported from the day of informed consent to the last date of contact for all participants.
Description: All enrolled participants who received at least 1 dose of study treatment. This study did not include a separate analysis of non-serious AEs therefore non-serious adverse events presented in this record include all adverse events reported during the study, not just non-serious events.
Arm/Group | Doxorubicin + Cyclophosphamide/Bevacizumab + Docetaxel
Serious Adverse Events (participants affected / at risk) | 13/72
Other Adverse Events (participants affected / at risk) | 71/72
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Doxorubicin + Cyclophosphamide/Bevacizumab + Docetaxel (N=72)
Febrile neutropaenia (Infections and infestations) | 6
Infection with normal absolute neutrophil count (ANC) or grade 1 or 2 neutrophils (Infections and infestations) | 1
Neutrophils/granulocytes (Blood and lymphatic system disorders) | 4
Mucositis/stomatitis (Gastrointestinal disorders) | 2
Vomiting (Gastrointestinal disorders) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Doxorubicin + Cyclophosphamide/Bevacizumab + Docetaxel (N=72)
Mucositis/stomatitis (Gastrointestinal disorders) | 43
Nausea (Gastrointestinal disorders) | 43
Vomiting (Gastrointestinal disorders) | 24
Diarrhoea (Gastrointestinal disorders) | 17
Constipation (Gastrointestinal disorders) | 14
Taste alteration (dysgeusia) (Gastrointestinal disorders) | 6
Anorexia (Gastrointestinal disorders) | 5
Heartburn/dyspepsia (Gastrointestinal disorders) | 6
Hair loss/alopecia (Skin and subcutaneous tissue disorders) | 36
Nail changes (Skin and subcutaneous tissue disorders) | 12
Rash: hand-foot skin reaction (Skin and subcutaneous tissue disorders) | 4
Other - not specified (Skin and subcutaneous tissue disorders) | 4
Fatigue (asthenia, lethargy, malaise) (General disorders) | 44
Fever (General disorders) | 14
Other - not specified (General disorders) | 5
Pain (General disorders) | 36
Neutrophils/granulocytes (Blood and lymphatic system disorders) | 10
Hemoglobin (Blood and lymphatic system disorders) | 5
Leukocytes (total WBC) (Blood and lymphatic system disorders) | 4
Infection with normal ANC or grade 1 or 2 neutrophils (Infections and infestations) | 17
Febrile neutropaenia (Infections and infestations) | 4
Allergic reaction/hypersensitivity (including drug fever) (Immune system disorders) | 14
Hemorrhage, pulmonary/upper respiratory (Respiratory, thoracic and mediastinal disorders) | 12
Watery eye (epiphora, tearing) (Eye disorders) | 7
Irregular menses (change from baseline) (Reproductive system and breast disorders) | 11
ALT, SGPT (serum glutamic pyruvic transaminase) (Metabolism and nutrition disorders) | 4
Cough (Respiratory, thoracic and mediastinal disorders) | 4
Other - not specified (Musculoskeletal and connective tissue disorders) | 6
Other - not specified (Renal and urinary disorders) | 5
Hypertension (Cardiac disorders) | 7
Hot flashes/flushes (Endocrine disorders) | 5
Flu-like syndrome (General disorders) | 9

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Study being conducted under this agreement is part of the Overall Study. Investigator is free to publish in reputable journals or to present at professional conferences the results of the Study, but only after the first publication or presentation that involves the Overall Study. The Sponsor may request the Confidential Information be deleted and/or the publication be postponed in order to protect the Sponsor's intellectual property rights.